CLINICAL TRIAL: NCT06983704
Title: Evaluation of Combined Bevacizumab-Mitomycin C Use During Ahmed Valve Revision in Recurrent Pediatric Glaucoma
Brief Title: Assessing Combined Bevacizumab-Mitomycin C Use During Ahmed Valve Revision in Recurrent Pediatric Glaucoma
Acronym: MMC glaucoma
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Ehab Mohamed Elsayed Mohamed Saad, Lecturer, Benha University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Bevacizumab-MMC; Benha University (Other: Al-Azhar University)
Record Dates: First submitted 2025-05-14; First posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2024-02

CONDITIONS: Pediatric Glaucoma
Keywords: Pediatric glaucoma; Ahmed valve; bevacizumab; mitomycin C
MeSH Terms: conditions — Hydrophthalmos | interventions — Bevacizumab

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Active Comparator): subconjunctival injection of bevacizumab was administered around the AGV plate using a 27-gauge needle
  Interventions: Procedure: AGV plate; Procedure: bevacizumab injection
- Group II (Active Comparator): AGV plate using a 27-gauge needle
  Interventions: Procedure: AGV plate

INTERVENTIONS:
Procedure: AGV plate — AGV plate using a 27-gauge needle
Procedure: bevacizumab injection — subconjunctival injection of bevacizumab
  Arms: Group I

SUMMARY:
To asess the efficacy and safety of combining subconjunctival bevacizumab with mitomycin C (MMC) during AGV revision surgery in pediatric patients with recurrent glaucoma.

DETAILED DESCRIPTION:
Recurrent pediatric glaucoma following Ahmed Glaucoma Valve (AGV) implantation presents a therapeutic challenge. This study evaluates the efficacy and safety of combining subconjunctival bevacizumab with mitomycin C (MMC) during AGV revision surgery in pediatric patients with recurrent glaucoma.

ELIGIBILITY:
Inclusion Criteria:

* children under 12 years with previous AGV implantation for primary congenital glaucoma

Exclusion Criteria:

* age >12 years, eyes with no light perception, and those with prior cyclodestructive procedures.

Max Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2024-02-09 (Actual); Primary Completion 2025-02-08 (Actual); Study Completion 2025-02-15 (Actual)

PRIMARY OUTCOMES:
surgical success | for 12 months
  IOP ≤ 21 mmHg and ≥ 5 mmHg without medications

CONTACTS AND LOCATIONS:
Locations (1):
- Al-Azhar University, Cairo, Egypt